CLINICAL TRIAL: NCT00960765
Title: Comparison Of Endotoxin Concentration And Intestinal Microbiologic Flora Before And After Roux-En-Y Gastric Bypass Or Gastric Banding Surgery In Morbidly Obese Patients With Type 2 Diabetes Mellitus
Brief Title: Endotoxin and Intestinal Flora Before and After Gastric Bypass or Banding in Diabetics
Status: Completed | Type: Observational
Sponsor: CPL Associates (Other)
Collaborators: Synergy Bariatrics (Unknown); Sisters of Charity Hospital (Unknown); The New York State Center of Excellence in Bioinformatics & Life Sciences (Other)
Responsible Party: Principal Investigator, Scott Monte, Program Director, CPL Associates
Other Study IDs: CPL200907A
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Obesity, Morbid; Diabetes Mellitus, Type 2; Gastric Bypass
Keywords: Type 2 Diabetes Mellitus; Gastric Bypass; Gastric Banding; Endotoxin
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, urine, stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Roux-En-Y Gastric Bypass
- Gastric Banding
- Sucessful Response to RYGB
- Failed Response to RYGB

SUMMARY:
This research project is designed to investigate endotoxin (a toxin present in the wall of certain kinds of bacteria) levels and the type of bacteria present in the intestine before and after Roux-en-Y gastric bypass or gastric banding surgery in patients that meet the classification for morbid obesity (body mass index >40 kg/m2) and type 2 diabetes. It is known that the type of bacteria present in the intestines of normal weight and obese individuals are different, and it is also known that people with obesity and type 2 diabetes have higher levels of endotoxin. It has been shown that the bacteria change over the long run after Roux-en-Y gastric bypass surgery, but the short-term effects are not known and the endotoxin levels after this procedure have never been studied.

DETAILED DESCRIPTION:
Evidence exists that (i) morbidly obese, T2D patients undergoing RYGB are highly likely to resolve T2D symptoms or dramatically reduce oral and/or insulin requirements, (ii) metabolic endotoxemia may incite the pathologic conditions of low-grade inflammation and subsequently insulin resistance, obesity and T2D, (iii) significant intestinal microbiologic flora differences exist between normal weight and obese/diabetic individuals, and (iv) RYGB alters long-term intestinal microbiologic flora. Therefore, it is logical to evaluate short- and long-term circulating endotoxin concentrations and intestinal microbiologic flora in context with weight loss and restoration of euglycemia to expand our knowledge of the mechanism of the benefits observed following RYGB.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age
* Morbid obesity (BMI > 40 kg/m2)
* Confirmed T2D diagnosis/date of onset

Exclusion Criteria:

* Age < 18 years of age
* BMI < 40 kg/m2
* Type 1 diabetes
* Chronic use of non-steroidal anti-inflammatory agents (NSAIDs)
* Chronic use of systemic corticosteroids
* Anticipated inability to maintain current statin, angiotensin converting enzyme inhibitor (ACEI), or angiotensin receptor blocking agent (ARB) regimen

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly obese (BMI > 40 kg/m2) patients with T2D
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2009-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Caruana, M.D., Principal Investigator — Synergy Bariatrics
Locations (2):
- United States (2):
  - Sisters of Charity Hospital, Buffalo, New York
  - Synergy Bariatrics, Williamsville, New York

REFERENCES:
- [Derived] Dandona P, Ghanim H, Monte SV, Caruana JA, Green K, Abuaysheh S, Lohano T, Schentag J, Dhindsa S, Chaudhuri A. Increase in the mediators of asthma in obesity and obesity with type 2 diabetes: reduction with weight loss. Obesity (Silver Spring). 2014 Feb;22(2):356-62. doi: 10.1002/oby.20524. Epub 2013 Sep 4. PMID 23804543
- [Derived] Ghanim H, Monte SV, Sia CL, Abuaysheh S, Green K, Caruana JA, Dandona P. Reduction in inflammation and the expression of amyloid precursor protein and other proteins related to Alzheimer's disease following gastric bypass surgery. J Clin Endocrinol Metab. 2012 Jul;97(7):E1197-201. doi: 10.1210/jc.2011-3284. Epub 2012 Apr 16. PMID 22508715